CLINICAL TRIAL: NCT04453982
Title: Is COVID-19 Transmitted Through Human Milk? Implications for Breastfeeding and Human Milk Banking-Study 1b
Status: Completed | Type: Observational
Sponsor: Deborah O'Connor (Other)
Collaborators: University of Toronto (Other); Sinai Health System (Other)
Responsible Party: Sponsor-Investigator, Deborah O'Connor, Scientist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 39373-b
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Sars-CoV2; Breastmilk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Human milk donors
  Interventions: Other: Human milk donors

INTERVENTIONS:
Other: Human milk donors — Human milk donors for the Rogers Hixon Ontario Human Milk Bank

SUMMARY:
The Canadian Paediatric Society recommends breastfeeding during COVID-19 infection. Human milk is the best form of infant nutrition providing significant protection against many illnesses for term and preterm infants. When mothers of hospitalized infants are unable to supply their milk, the recommended supplement is human donor milk. The impact of a pandemic on human milk banking is unknown. This study seeks to address this public health issue. Donor milk will be collected from the Rogers Hixon Ontario Human Milk Bank at Sinai Health System in Toronto. Samples will be analyzed for the COVID-19 virus specific nucleic acid and antibody in real-time and results will be immediately disseminated to relevant organizations to inform local, national and international guidelines surrounding donor milk banking to protect the health of infants.

ELIGIBILITY:
Inclusion Criteria:

- Human milk donor for the Rogers Hixon Ontario Human Milk Bank

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 in breastmilk | 2 months
  To describe the prevalence of human milk donations received at the Ontario Human Milk Bank that test positive for SARS-CoV-2
Prevalence of SARS-CoV-2 antibody in breastmilk | 2 months
  To describe the prevalence of human milk donations received at the Ontario Human Milk Bank with antibodies for SARS-CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Health System, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ismail S, Unger S, Budylowski P, Poutanen S, Yau Y, Jenkins C, Anwer S, Christie-Holmes N, Kiss A, Mazzulli T, Johnstone J, McGeer A, Whittle W, Parvez B, Gray-Owen SD, Stone D, O'Connor DL. SARS-CoV-2 antibodies and their neutralizing capacity against live virus in human milk after COVID-19 infection and vaccination: prospective cohort studies. Am J Clin Nutr. 2024 Feb;119(2):485-495. doi: 10.1016/j.ajcnut.2023.10.008. Epub 2023 Dec 14. PMID 38309831